CLINICAL TRIAL: NCT06909695
Title: Influences of Long-acting Reversible Contraceptives on Iron Status and Physiological Responses to Extreme Environments in Women
Status: Recruiting | Type: Observational
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 24-19
Record Dates: First submitted 2024-10-04; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Contraception; Iron Deficiencies
MeSH Terms: conditions — Iron Deficiencies | interventions — Blood Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples, without DNA, for analysis of biomarkers of environmental stress
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SARC: Control group utilizing short-acting reversible contraceptives (i.e. combined oral contraceptives tested only in the active pill phase or transdermal patch)
  Interventions: Other: Blood volume and environmental testing
- LARC users: Users of hormonal long-acting reversible contraceptives (LARCs) (e.g. hormonal IUDs, hormonal subcutaneous implants)
  Interventions: Other: Blood volume and environmental testing

INTERVENTIONS:
Other: Blood volume and environmental testing — Testing blood volume measures, iron stores, and physiological responses to acute environmental exposures of heat, cold, and high-altitude (each environment independently)

SUMMARY:
Over recent years, military service women have shown increasing interest in utilizing long-acting reversible contraceptives (LARCs; i.e., implants or intrauterine devices, IUDs). While clinically, LARC have been proven safe and effective at preventing pregnancy & decreasing menstrual symptoms, it is unclear what impact this type of contraceptive may have on physiological responses to extreme environments (heat, cold and high altitude). Additionally, iron deficiency and iron deficiency anemia are prevalent in U.S. military women which likely affect health and performance. There is evidence to suggest that the prevalence of iron deficiency and iron deficiency anemia is lower in women utilizing LARCs, which preserve iron stores, likely due to reduced menstrual blood loss that compounds with each cycle over the course of months. Due to the increasing interest in the utilization of LARCs it is important to understand what, if any, impact these methods of contraception may have on a female Soldier's physiological responses.

The overall goal of the present study is to characterize iron status and physiological responses (including but not limited to sweating, skin blood flow, ventilation, and heart rate) to extreme environmental stressors of heat, cold and high altitude (i.e. hypobaric hypoxia) in women utilizing LARCs. Up to thirty-three individuals (n=18 LARCs, n=15 monophasic oral contraceptives) will complete testing visits separated by at least 48 hours for environmental testing visits. During heat stress testing, measures of core body temperature, skin temperature, and sweat rate will be measured during a standardized protocol in hot, humid conditions. During cold stress, measures of body core temperature, metabolic heat production, skin blood flow and temperature (at both distal extremity and proximal body sites) will be assessed in order to better quantify the impact of exogenous sex hormones via LARCs and OCs in volunteers exposed to the cold. Measurements will be obtained during a standardized protocol in cold air (~90 min; 10°C). For altitude, cardiopulmonary responses will be assessed during rest and exercise during an acute altitude exposure (4300m). Blood samples will be collected throughout the investigation in order to quantify sex hormone concentrations, iron status, and inflammatory biomarkers in response to environmental stressors. The investigators will also utilize laboratory tests (i.e., carbon monoxide (CO) rebreathing technique) and collect blood samples to quantity iron stores in these groups of women. To characterize iron status, the Soldier Performance Health and Readiness (SPHERE) epidemiological data repository will be utilized to quantify the prevalence of iron deficiency and iron deficient anemia diagnoses between women using LARCs and women not utilizing LARCs.

ELIGIBILITY:
Inclusion Criteria:

* • Females, age 18-40 y

  * Females taking monophasic oral contraceptives or utilizing implantable contraception (intrauterine device, implantable bar) for at least one year, and be at least one year removed from the removal end point (e.g. before year 4 for a 5-year IUD)
  * In good health as determined by OMSO (Office of Medical Support and Oversight)
  * Passed most recent Army Combat Fitness Test (ACFT) (military volunteers only) or exercise at least 2 times per week (civilian volunteers)
  * Willing to not drink alcoholic beverages for 24 hours before each testing session
  * Willing to not consume caffeine 12 hours prior to any testing sessions
  * Willing to refrain from any exercise and additional moderate to strenuous physical activity 24 hours prior to testing
  * Willing to stay and exercise in an altitude chamber (the size of a dorm room) for ~6 hours
  * Supervisor approval for federal civilian employees and non-HRV active-duty military personnel stationed at NSSC.

Exclusion Criteria:

* • Females who are pregnant, planning to become pregnant during the study, or breastfeeding.

  * Taking prescription, over the counter medication, or dietary supplements, other than a contraceptive (unless approved by OMSO and Principal Investigator (PI))
  * Tobacco or nicotine users, or anyone who has used tobacco or nicotine within the last four months
  * Physical problems/injuries (e.g., current stress fractures, musculoskeletal strains) that would affect walking or running on a treadmill
  * Allergy to skin adhesive
  * Heart, lung, kidney, muscle, endocrine, or nerve disorder(s) as determined by OMSO
  * History of heat intolerance or orthostatic intolerance
  * Diagnosed and/or treated for fluid/electrolyte imbalance within the last 30 days
  * History of obstructive disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis.
  * Scheduled MRI within 2 weeks after completing a heat or cold test
  * Actively dieting with the intent to lose weight
  * History of cold injuries of any severity (e.g., frostbite, trench foot, chilblains).
  * Raynaud's syndrome
  * Cold-induced asthma/bronchospasm
  * Not willing to have small areas of skin on the body shaved (if deemed necessary for attachment of study instrumentation)
  * Born at altitudes greater than 2,100 m (7,000 ft) (e.g., Mexico City, Mexico)
  * Living in areas that are more than 1,200 m (4,000 ft) (e.g., Colorado Springs, CO) or have traveled to areas that are more than 1,200 m for five days or more within the last 2 months
  * Prior diagnosis of High Altitude Pulmonary Edema (HAPE) or High Altitude Cerebral Edema (HACE)
  * Abnormal blood count in accordance with OMSO - Normal Hb women: 11.1-15.9 g·dL-1 or Normal Hct women: 34.0-48%, or presence of abnormal blood chemicals (hemoglobin S or Sickle Cell Trait)
  * History of pneumothorax
  * History of hypertension
  * Blood donation within 8 weeks of beginning the study
  * Any recent (within 4-6 weeks) and or expected history of prolonged periods of immobility or limited activity (including recent or upcoming surgery)
  * Evidence of apnea or sleeping disorder (narcolepsy, insomnia, etc.)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity and the inclusion criteria of utilizing either combined oral contraceptives or long-acting reversible contraceptives
Study Population: The proposed population will be healthy and active women between the ages of 18-40. This population is suitable for the purpose of this investigation since they are the most militarily relevant population (i.e., representative of the U.S. Army active duty population).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Iron status | upon initial visit
  Iron stores as measured by ferritin levels
Ventilation | intermittently throughout high-altitude trial (5 timepoints overall over ~6-7 hours)
  ventilatory response to high altitude exposure at rest and during exercise
Thermoregulation in the heat - core temperature | measured intermittently throughout trial (at least every 5 minutes) for 2 hour exposure
  Measure of core temperature
Thermoregulation in the cold - skin blood flow | measured intermittently throughout cold trial (at least every 5 minutes) for 2 hour exposure
  Measure of thermoregulation during resting cold stress to include skin blood flow
Thermoregulation in the heat - skin temperature | measured intermittently throughout trial (at least every 5 minutes) for 2 hour exposure
Thermoregulation in the heat - sweating rate | Only measured during heat stress visit, at one timepoint immediately after exercise on heat stress visit (post-exercise, within 10-20 minutes)
  Calculated from pre- and post-nude body mass corrected for fluid consumed and urine produced
Thermoregulation in the cold - core temperature | measured intermittently throughout cold trial (approximately every 5-10 min) for 2 hour exposure
Thermoregulation in the cold - skin blood flow | measured intermittently throughout cold trial (approximately every 5-10 minutes) for 2 hour exposure

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Giersch, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No